CLINICAL TRIAL: NCT04082715
Title: Transition From Acute to Chronic Back Pain : Effect of L-dopa,Gender,and Associated Brain Plasticity
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: we don't have enough research funding.
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-05-105
Record Dates: First submitted 2019-08-06; First posted 2019-09-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Chronic Back Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Carbidopa; Levodopa; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- carbidopa/levodopa+celecoxib (Experimental): carbidopa/levodopa+celecoxib treatments will be effective.
  Interventions: Drug: carbidopa/levodopa and celecoxib
- placebo1+celecoxib (Placebo Comparator): A placebo comparator for carbidopa/levodopa+celecoxib .
  Interventions: Drug: placebo1 and celecoxib
- placebo1+placebo2 (Placebo Comparator): A placebo comparator for carbidopa/levodopa+celecoxib and placebo1+celecoxib.
  Interventions: Drug: placebo1 and placebo2

INTERVENTIONS:
Drug: carbidopa/levodopa and celecoxib — Every patient of this arm will get one bottle of carbidopa/levodopa and one bottle of celecoxib. At treatment initiation, Carbidopa/Levodopa will be taken once daily for 3 days, then twice daily for 3 days, and then thrice daily over one week and then continue on that dose for the duration of the treatment period (12 weeks total). At the last treatment visit (end of the treatment period), patients will begin tapering off the medication as follows. S/he will start with carbidopa/levodopa twice daily for 3 days and then once daily for 3 days before discontinuing it completely.Celecoxib will remain constant once daily for patients of this arm throughout the treatment period, but it will not be given during the tapering down at the end of the treatment period(12 weeks total).
  Arms: carbidopa/levodopa+celecoxib
Drug: placebo1 and celecoxib — Every patient of this arm will get one bottle of placebo1 and one bottle of celecoxib. At treatment initiation, placebo1 will be taken once daily for 3 days, then twice daily for 3 days, and then thrice daily over one week and then continue on that dose for the duration of the treatment period (12 weeks total). At the last treatment visit (end of the treatment period), patients will begin tapering off the medication as follows. S/he will start with placebo1 twice daily for 3 days and then once daily for 3 days before discontinuing it completely. Celecoxib will remain constant once daily for patients of this arm throughout the treatment period, but it will not be given during the tapering down at the end of the treatment period(12 weeks total).
  Arms: placebo1+celecoxib
Drug: placebo1 and placebo2 — Every patient of this arm will get one bottle of placebo1 and one bottle of placebo2. At treatment initiation, placebo1 will be taken once daily for 3 days, then twice daily for 3 days, and then thrice daily over one week and then continue on that dose for the duration of the treatment period (12 weeks total). At the last treatment visit (end of the treatment period), patients will begin tapering off the medication as follows. S/he will start with placebo1 twice daily for 3 days and then once daily for 3 days before discontinuing it completely. placebo2 will remain constant once daily for patients of this arm throughout the treatment period, but it will not be given during the tapering down at the end of the treatment period(12 weeks total).
  Arms: placebo1+placebo2

SUMMARY:
This is a 6-month double-blinded, randomized, placebo-controlled clinical trial of pharmacological treatment (carbidopa/levodopa and celecoxib) for acute/subacute back pain. All eligible patients will be randomly assigned to 3 different group and receive a 12-week treatment of "carbidopa/levodopa+celecoxib ", of "placebo+celecoxib", and of "placebo+placebo". In addition, all participants will be MRI-scanned twice and assessed daily with a mobile app for pan, mood, and behavior.

DETAILED DESCRIPTION:
This is a 6-month double-blinded, randomized, placebo-controlled clinical trial of pharmacological treatment for acute/subacute back pain (carbidopa/levodopa and celecoxib).The dosage of carbidopa/levodopa is 25/100mg.After screening, all eligible patients will be randomly assigned to 3 different groups, with each receives a 12-week treatment of "carbidopa/levodopa+celecoxib (LDP+CLX)", of "placebo+celecoxib (PLC+CLX)", and of "placebo+placebo (PLC+PLC)". For each group, a subsequent 12-week follow-up efficacy evaluation will be conducted by telephone .At the end of the 24-week study, we will understand the durability of the treatment. During the drug treatment period for pain, all participants should return to the clinical follow-up center on week 0, 2, 6 and 12 to assess pain condition, properness of treatment and side effects .In the 24-week study of drug treatment and after treatment follow-up, pain and safety assessments will be conducted by telephone, at week 9, 16, and 20.In addition, all participants will be assessed daily with a mobile app for pain, mood and behavior.Participants will be scanned for brain structure images (T1), resting functional images (RS-fMRI) and diffusion tensor images (DTI) at the second follow-up visit (week 0) and at the end of study (week 24).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* New onset subacute or acute back pain (< 6 months' duration, no back pain for 3 months before the new onset)
* Signs and symptoms: positive straight leg raising test with dermatomal radiation and/or myotomal weakness and/or reflex asymmetry, pain must radiate into buttock or below
* Average reported pain intensity from App greater than 4/10 during the first week
* MUST be able to undergo MRI procedures (no pacemaker, any metal implants)

Exclusion Criteria:

* Previous (distinct) episodes of back pain onset (more than 3 distinct episodes of back pain lasting for a total of more than 4 weeks) in the previous year;
* Evidence of acute vertebral fracture;
* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills;
* Symptoms of neuropathy due to diabetes Type I or Type II;
* Chronic neurologic conditions, including Parkinson's disease, Alzheimer's disease, and other conditions associated with dementia;
* Significant other medical diseases such as congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy;
* History of glaucoma or narrow angle glaucoma;
* Presence of undiagnosed skin lesions or history of melanoma;
* Presence of severe cardiovascular or pulmonary disease, bronchial asthma, renal, hepatic or endocrine disease;
* History of myocardial infarction with residual cardiac arrhythmia;
* History of gastrointestinal bleeding or peptic ulcer;
* Diagnosis of current depression (assessed via BDI, total > 28 are excluded) or psychiatric disorder requiring treatment, or such a diagnosis in the previous 6 months;
* Use of therapeutic doses of antidepressant medications (i.e., tricyclic antidepressants, SSRIs, SNRIs; low doses used only in the evening for sleep will be allowed if dose is not changed;
* Current use of recreational drugs or recent history of alcohol abuse (pattern of drinking having social, financial or physical consequences) or drug abuse (urine screening);
* Current use of cannabinoids (4 participants tested positive; 3 completed the study, in these blood test at the end of the study confirmed cannabinoid use; excluding these subjects does not importantly alter results, see below);
* High dose opioid prophylaxis, defined as > 50mg morphine equivalent/day;
* Use of MAOIs, currently or within the past 2 weeks;
* Prior use of levodopa;
* Use of any of the following drugs: bromocryptine, linezolid, metoclopramide, phenothiazines, promethazine/codeine, isoniazid, rifampin, pyrazinamide;
* Oral iron supplementation;
* Currently taking levodopa or dopaminergic drugs
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions
* For those receiving MRI: intra-axial implants (e.g. spinal cord stimulators or pumps), all exclusion criteria for MR safety: any metallic implants, pacemaker, brain or skull abnormalities, tattoos on large body parts, and claustrophobia;
* Pregnancy or inability to use an effective method of birth control in sexually active men and women while taking the study drug and for one week thereafter. Barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUD's), hormonal contraceptives, oral contraceptive pills, surgical sterilization, and complete abstinence are examples of effective methods of contraception;
* Following laboratory abnormalities: liver function tests (SGOT/SGPT) greater than twice the upper limit of normal; unexplained anemia (Hgb 13.5 to 17.5 g/dL for men, 12.0 to 15.5g/dL for women); evidence of renal insufficiency (creatinine >upper limit of normal) or any other abnormality that the principal investigator feels puts the participant at risk during the study. A blood re-test could occur for all enrolled subjects within one month of the first blood draw due to potential risk for renal impairment with NSAIDs at this dosage;
* History of chronic opioid use for pain management;
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk.
* Contraindications to use of study product, based on any of the following:
* Hypersensitivity to carbidopa/levodopa or other constituents of the carbidopa/levodopa capsules;
* Hypersensitivity to lactose or other constituents of the placebo capsules;
* Hypersensitivity to naproxen or other constituents of the celecoxib capsules;
* Hypersensitivity to acetaminophen or other constituents of the acetaminophen tablets;
* Taking concomitant medication which may be adversely affected by omeprazole to a degree that alters subject's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity of subjects | Baseline, 12th week, 24th week
  Numeric Rating Scale is an 11-point numerical rating scale used to measure pain intensity, the minimum score is 0 and maximum score is 10,the number 0 presents no pain, and number 10 presents the worst imaginable pain.The higher value represent a worse outcome.

SECONDARY OUTCOMES:
Brain regional gray matter density of subjects | Baseline, 24th week
  All the subjects will be scanned by MRI for contrasting anatomical brain image, and the brain regional gray matter density will be calculated from the contrasting anatomical image.
Brain functional connectivity strength | Baseline, 24th week
  All the subjects will be scanned by MRI for functional brain images, and the brain functional connectivity strengths will be calculated from the functional brain images, with number 1 presents the maximum positive connectivity between two different brain regions, number -1 presents maximum negative connectivity, and number 0 presents 0 connectivity.

OTHER OUTCOMES:
Sensory and affective components of pain of subjects | Baseline, 12th week, 24th week
  The scores of The McGill Pain Questionnaire is a well-validated pain measure with sensory and affective components of pain.
  The McGill Pain Questionnaire descriptors fall into two major groups: Sensory; Affective. The lowest possible score for each question is 0, the highest possible score for each question is 3, the higher value represent a worse outcome.
  Sensory (sections 1-11): The scores can range from 0 to 33. Affective (sections 12-15): The scores can range from 0 to 12.
Positive and negative mood affect of subjects | Baseline, 12th week, 24th week
  The Positive and Negative Affect Schedule has two mood scales, one measuring positive affect and the other measuring negative affect .The lowest possible score for each question is 1, the highest possible score for each question is 5.
  Positive Affect Schedule(sections 1,3,5,9,10,12,14,16,17,19): Scores can range from 10 to 50, with higher scores representing higher levels of positive affect.
  Negative Affect Score(sections 2,4,6,7,8,11,13,15,18,20): Scores can range from 10 to 50, with lower scores representing lower levels of negative affect.
The severity of depression of subjects | Baseline, 12th week, 24th week
  Beck's Depression Index add up the score for each of the 21 questions . The lowest possible score for each question is 0, the highest possible score for each question is 3. The possible total scores can range from 0 to 63, the higher value represent a worse depression.
Individual pain sensitivity of subjects | Baseline, 12th week, 24th week
  Pain Sensitivity Questionnaire (PSQ)is a 11-point, 17-item instrument used to assess individual pain sensitivity.
  PSQ-minor and PSQ-moderate were two subscales corresponding to mildly painful and moderately painful situation respectively.
  PSQ-minor(sections 3,6,7,10-12,14): the lowest possible score for each question is 0 the highest possible score for each question is 10. Scores can range from 0 to 70.
  PSQ-moderate(sections 1,2,4,8,15-17): the lowest possible score for each question is 0 the highest possible score for each question is 10. Scores can range from 0 to 70.
  The higher value represent more sensitive.
Thoughts or feelings on past pain experience of subjects | Baseline, 12th week, 24th week
  The Pain Catastrophizing Scale is a 5-point instrument to assess 13 thoughts or feelings on past pain experience.
  The Pain Catastrophizing Scale yields three sub-scale scores assessing rumination, magnification , and helplessness. The lowest possible score for each question is 0 the highest possible score for each question is 4. The higher value represent a worse outcome.
  Rumination(sections 8-11): The total score of the four items can range from 0 to 16.
  Magnification(sections 6,7,13):The total score of the three items can range from 0 to 12.
  Helplessness(sections 1-5,12): The total score of the six items can range from 0 to 24.
Fear and anxiety responses specific to pain of subjects | Baseline, 12th week, 24th week
  Pain Anxiety Symptom Scale measures fear and anxiety responses specific to pain. It has 13 questions consisted of four aspects of pain-related anxiety.
  Cognitive suffering(sections 1-5): the lowest possible score for each question is 0 the highest possible score for each question is 5. Scores can range from 0 to 25. Escape-avoidance behaviors(sections 6-10): the lowest possible score for each question is 0 the highest possible score for each question is 5. Scores can range from 0 to 25.
  Fear of pain(sections 11-15): the lowest possible score for each question is 0 the highest possible score for each question is 5. Scores can range from 0 to 25. Physiological symptoms of anxiety(sections 16-20): the lowest possible score for each question is 0 the highest possible score for each question is 5. Scores can range from 0 to 25.
  The higher value represent a worse anxiety.
Physical impairment in relation to pain of subjects | Baseline, 12th week, 24th week
  Pain Disability Index has 11-point, where 0 corresponds to no disability and 10 indicates worst disability.The lowest possible score for each question is 0(best), the highest possible score for each question is 10(worst). the total score of the seven items can range from 0 to 70, the higher value represent a worse disability.

CONTACTS AND LOCATIONS:
Overall Officials: BinBin Wu, doctor, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China